IRAS ID: 290193

Reference Number: 1

Date: 26/04/2022 Version Number: 3

To Examine the Effectiveness of Physical Activity, Quality of Life and Hospital Anxiety and Depression Outcomes in Cardiovascular Patients

Using Either Traditional, Web-based or a Combined Cardiac rehabilitation Programme.

NCT 05326529

26th April 2022

IRAS ID: 290193

Reference Number: 1 Date: 26/04/2022 Version Number: 3



Centre Number: Study Number:

Participant Identification Number for this trial:

## **CONSENT FORM**

**Title of Project:** To examine the effectiveness of Physical Activity, Quality of Life and Hospital Anxiety and Depression outcomes in Cardiovascular patients using an internet-based Cardiac Rehabilitation application compared with a conventional Cardiac Rehabilitation programme or a combination of both.

| with a | a conventional Cardi | ac Rehabilitation programme or a d | combination of both. | |
|---|---|---|---|---|
| Name | e of Researcher: Ch | narlotte Smith and Francesca D'An | gelo | Please initial box |
| 1. | I confirm that I have read the information sheet dated (25/04/2022) for the above study. I have had the opportunity to consider the information, ask questions and had these answered satisfactorily. | | | nave |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | | | |
| 3. | I understand that relevant sections of my medical notes and data collected during the study, may be looked at by other individuals within the cardiac rehabilitation team, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | | |
| 4. | I agree my GP may be contacted for support if the research team has concerns about my mental health and/or safety. | | | |
| 5. | 5. I agree to take part in the above study. | | | |
| 6. | I would like to rece | ive a copy of the study results. | Yes | No |
| Name | e of Participant | Date | Signature | |
| Name of Person seeking consent | | Date | Signature | |